CLINICAL TRIAL: NCT00634569
Title: Evaluation of the Efficacy and Safety of Flebogamma 5% DIF [Immune Globulin Intravenous (Human)] for Replacement Therapy in Pediatric Subjects With Primary Immunodeficiency Diseases.
Brief Title: Safety and Efficacy Study of Flebogamma 5% DIF IGIV in Pediatric Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Organization: Grifols Biologicals, LLC (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IG-0705
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Results first posted 2016-12-08 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-12

CONDITIONS: Primary Immune Deficiency Disease
Keywords: CVID, XLA, hyper IgM syndrome, Wiskott-Aldrich Syndrome
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Bruton type agammaglobulinemia; Hyper-IgM Immunodeficiency Syndrome; Wiskott-Aldrich Syndrome | interventions — gamma-Globulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Flebogamma 5% DIF (Experimental)
  Interventions: Biological: Flebogamma 5% DIF

INTERVENTIONS:
Biological: Flebogamma 5% DIF — Intravenous Immune Globulin (Human)

SUMMARY:
This is a multi-center, open-label study to assess the efficacy and safety of Flebogamma 5% DIF in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* The subject is between 2 and 16 years old, of either sex, belonging to any ethnic group, and above a minimum weight of 10 kg (this weight is based on the amount of blood required for testing).
* The subject has a primary immunodeficiency disease, (e.g., common variable immunodeficiency, X-linked and autosomal forms of agammaglobulinemia, hyper-IgM syndrome, Wiskott-Aldrich Syndrome).
* The subject has been receiving licensed IGIV replacement therapy at a dose that has not changed by + 50% of the mean dose on a mg/kg basis for at least 3 months before study entry and has maintained a trough level at least 300 mg/dL above baseline serum IgG levels.
* Trough levels of IgG, dose of IGIV, and treatment intervals for the last 2 consecutive routine IGIV treatments must be documented for each subject before the first infusion in this study can be administered.
* If a subject is an adolescent female (> 12 years of age) who is or becomes sexually active, she must have a negative result on a pregnancy test (HCG-based assay).
* The subject, if old enough (generally 6 years to 16) has signed an informed Child Assent form and the subject's parent or legal guardian has signed an informed consent form, both approved by the Institutional Review Board.

Exclusion Criteria:

* Adult patient (> 17 years old).
* The subject has a history of any severe anaphylactic reaction to blood or any blood-derived product.
* The subject is known to be intolerant to any component of the products, such as sorbitol (i.e., intolerance to fructose).
* The subject has selective IgA deficiency or has demonstrable antibodies to IgA.
* The subject is currently receiving, or has received, any investigational agent within the prior 3 months.
* The subject has been exposed to blood or any blood product or derivative within the last 6 months, other than a commercially available IGIV.
* The adolescent subject is pregnant or is nursing.
* The subject, at screening, has levels greater than 2.5 times the upper limit of normal as defined at the central laboratory for pediatric patients of any of the following:

  * ALT
  * AST
  * LDH
* The subject has a severe pre-existing renal impairment (defined by serum creatinine greater than 2 times the ULN or BUN greater than 2.5 times the ULN for that laboratory, or any subject who is on dialysis) or any history of acute renal failure.
* The subject has a history of DVT or thrombotic complications of IGIV therapy.
* The subject suffers from any acute or chronic medical condition (e.g., renal disease or predisposing conditions for renal disease, coronary artery disease, or protein losing state) that, in the opinion of the Investigator, may interfere with the conduct of the study.
* The subject has an acquired medical condition such as lymphocytic leukemia, chronic or recurrent neutropenia (ANC less than 1000), or AIDS known to cause secondary immune deficiency, or is s/p hematopoetic stem cell transplantation.
* The subject is receiving the following medication:

  * Systemic corticosteroids (long-term, i.e., not intermittent or burst, daily, > 1 mg of prednisone equivalent/kg/day). Topical steroids (ie- nasal, inhaled for asthma, and/or skin preparations for eczema) are not exclusionary.
  * Immunosuppressive drugs
  * Immunomodulatory drugs
* The subject has non-controlled arterial hypertension (systolic blood pressure > 160 mm Hg and/or diastolic blood pressure > 100 mm Hg).
* The subject has anemia (hemoglobin < 10 g/dL) at screening.
* The subject and/or parent/legal guardian of the subject is unlikely to adhere to the protocol requirements of the study or is likely to be uncooperative or unable to provide from the patient a storage serum sample at the screening visit. (Please note, a pre-treatment serum sample to be stored at -94° F (-70º C) for possible future testing is absolutely required).

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2008-05; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ballow, MD, Principal Investigator — Children's Hospital of Buffalo
Locations (7):
- United States (7):
  - University of South Florida, St. Petersburg, Florida
  - Family Allergy & Asthma Center, PC, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - The Allergy and Asthma Center, Fort Wayne, Indiana
  - The Children's Hospital of Buffalo, Buffalo, New York
  - Pennsylvania State University, Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital and Regional Medial Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- 21-day Dosing: IGIV given every 21-days (225-600 mg/kg)
- 28-day Dosing: IGIV given every 28-days (300-800 mg/kg)
Period: Overall Study
Arm/Group | 21-day Dosing | 28-day Dosing
Started | 14 | 10
Completed | 14 | 5
Not Completed | 0 | 5
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 21-day Dosing | 28-day Dosing | Total
Number analyzed (Participants) | 14 | 10 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.6 (4.3) | 9.7 (4.9) | 9.0 (4.53)
Gender [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 10 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 14 | 8 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Serious Bacterial Infections.
Description: Total number of Bacterial pneumonia, bacteremia or sepsis, osteomyelitis/septic arthritis, visceral abscess or bacterial meningitis
Time Frame: 12 months
Measure: Number; unit: Total serious bacterial infections
Arm/Group | 21-day Dosing | 28-day Dosing
Number analyzed (Participants) | 14 | 10
Total serious bacterial infections | 1 | 0

2. Secondary Outcome: Days of School/Usual Activities Missed Per Year
Description: Mean Days of school/usual activities missed per subject/year
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Days
Groups:
- All Subjects: Intent-to-treat population
Arm/Group | All Subjects
Number analyzed (Participants) | 24
Days | 2.0 (3.33)

3. Secondary Outcome: Days of Hospitalization Per Year
Description: Mean Days of hospitalization per subject/year
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | All Subjects
Number analyzed (Participants) | 24
Days | 0.2 (1.04)

4. Secondary Outcome: Number of Visits to Physician/ER Room for Acute Problems
Description: Mean Number of visits to physician/ER room for acute problems
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | All Subjects
Number analyzed (Participants) | 24
Visits | 0 (0.0)

5. Secondary Outcome: Other Infections Documented by Fever and Physical Exam or Positive Radiograph.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Number of other infections
Arm/Group | All Subjects
Number analyzed (Participants) | 24
Number of other infections | 0 (0.0)

6. Secondary Outcome: Number of Infectious Episodes Per Year
Description: Mean Number of infectious episodes per subject/year
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Infectious episodes
Arm/Group | All Subjects
Number analyzed (Participants) | 24
Infectious episodes | 0.9 (1.44)

7. Secondary Outcome: Number of Days on Antibiotics (Prophylactic and Therapeutic).
Description: Median Combined number of days on prophylactic and therapeutic antibiotics
Time Frame: 12 months
Measure: Median (Standard Deviation); unit: Days
Arm/Group | All Subjects
Number analyzed (Participants) | 24
Days | 72 (150.45)

8. Secondary Outcome: Number of Adverse Events
Description: Total Number of Adverse Events
Time Frame: 12 months
Measure: Number; unit: All Adverse Events
Arm/Group | All Subjects
Number analyzed (Participants) | 24
All Adverse Events | 159

ADVERSE EVENTS:
Time Frame: 1 year
Description: Systematic temporal assessment of AEs (by vital sign measurement up to 72 hours post-infusion) occurring over 1 year
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 1/24
Other Adverse Events (participants affected / at risk) | 15/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=24)
Cellulitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Femoral neck fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=24)
Headache (General disorders) | 10 (31)
Diastolic hypotension (Nervous system disorders) | 5 (20)
Pyrexia (Infections and infestations) | 7 (19)
Hypotension (Nervous system disorders) | 6 (19)
Tachycardia (Cardiac disorders) | 6 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No